CLINICAL TRIAL: NCT00457132
Title: Dynamic Wedging: A Novel Treatment for Knee Osteoarthritis
Brief Title: The Effect of Neuromuscular Training on Osteoarthritis: A Comparative Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44/05
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; WOMAC; ALF; Wedging
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APOS biomechanical gait system

SUMMARY:
Context: The many treatments and devices developed to unload the diseased articular surface in knee osteoarthritis have provided limited solutions. A novel biomechanical device comprising of four individually calibrated elements attached onto foot-worn platforms was recently developed. This device is capable of such unloading during standing and walking, simultaneously strengthening dynamic stabilizers and training neuromuscular control by controlled biomechanical perturbations.

Objective: To asses the effectiveness of this device in reducing pain and improving function in patients with knee osteoarthritis.

Design and Setting: Randomized, controlled and double blind prospective trial, conducted from September 2005 to February 2006, in the Department of Orthopedics, Asaf Harofeh Medical Center (Zerifin, Israel).

Patients: Sixty-one patients with diagnosed knee osteoarthritis who self-reported moderate-to-severe level pain.

Interventions: Patients were randomly assigned into active and control groups and underwent 8 weeks of treatment. The active group was treated with the device and its four biomechanical elements that had been individually calibrated to accommodate a pain-free joint alignment. The control group was treated with the device's platforms without the biomechanical elements.

Primary Outcome Measures: The patients were evaluated three times during the study: at baseline, after 4 weeks and at the 8 week endpoint. Primary outcomes were the Western Ontario and McMaster Osteoarthritis Index (WOMAC) and the Aggregated Locomotor Function (ALF) assessment.

DETAILED DESCRIPTION:
The Biomechanical System The biomechanical system is a biomechanical device (US Patent No. 6,979,287) combined with a treatment methodology (US Patent No. 7,101,330). The device is calibrated for the individual patient according to pathology and motion characteristics. Appropriate calibration is defined as bringing the damaged joint to a biomechanical alignment that minimizes/eliminates pain by shifting and/or changing the applied forces and, consequently, altering pressure distribution within the joint. Together with the biomechanical perturbation applied through all phases of the step-cycle (i.e. initial contact, mid-stance and toe-off), this enables home-based, dynamic, functional and repetitive training to strengthen dynamic stabilizers and improve neuromuscular control.

The device consists of two half spherical-shaped biomechanical elements attached to each of the patient's feet. One is located under the hindfoot region and the other is located under the forefoot region. The elements are available in different degrees of resilience and convexity, and are attached to the patient's foot using a platform in the form of a shoe. The platform is equipped with a specially designed sole, which consists of two mounting rails to enable flexible positioning of each element under each region.

A specific level of "unloading" under a specific level of perturbation is required for controlling pain in the affected compartment while reducing excessive loads of soft tissue structures. Primary guidelines for calibration dictate the choice of resilience, convexity and the position of each element. For example, in a genu-varus deformity the elements are positioned under the neutral axis of the patient's leg. The element under the hindfoot is further translated laterally to the longitudinal axis of the patient's leg in order to apply wedging, while the element under the forefoot is further translated medially to reduce the tension applied by soft tissue in the medial compartment, and to decrease adduction moment. When required, further soft tissue tension and/or pressure can be decreased by adding plantar flexion and/or forward translation of the hindfoot element.

Pain and motion instability are periodically evaluated to determine whether recalibration is required.

Treatment (Active) Protocol The device was calibrated for each patient after baseline assessment. Then, treatment was initiated and continued daily for a period of 8 weeks, during which the device was again calibrated, as necessary, after the first, third and sixth week. Patients were instructed to follow a treatment protocol which was based on walking during activities of daily living and started with 10 minutes of indoor walking each day during the first week and gradually increased to 30 minutes of daily outdoor walking in the last week. Other than that, they were told to continue their daily activities wearing their regular footwear. They were also instructed not to ingest any pain relief medication, non-steroidal anti-inflammatory drugs or food supplements except for the acetaminophen tablets (unmarked) that had been given to them at study entry to be taken when needed. The consumption of acetaminophen or any other medication was monitored during each assessment.

Control Protocol Patients in the control group were fitted with a platform which was identical in appearance but had a regular sole and did not include the biomechanical elements. They were instructed to follow the same treatment protocol as the active group and not to ingest any medication or food supplement apart from the unmarked acetaminophen tablets that had been given to them.

Assessment We tested the clinical efficacy of a device designed for reducing pain and improving function in knee osteoarthritis patients by means of the self-reported Western Ontario and McMaster Osteoarthritis Index (WOMAC) and the measured aggregated locomotor function (ALF). The WOMAC is composed of a 5 items pain scale, a 2 items stiffness scale and a 17 items function scale. All 24 items are rated by the patients on a visual-analogue-scale (in cm) from 0 (no symptoms/limitations) to 10 (maximal symptoms/limitations). The ALF scale is a sum of mean timed score (seconds) of three locomotor functions: time taken to walk 8 meters, time taken to accent and decent 7 stairs and time taken to transfer from sitting to standing. The patients were evaluated three times during the study: at baseline, after 4 weeks and at the 8 week endpoint. Measurements were made with the patients barefooted as required by the outcome protocol.

To ensure our ability to detect clinically significant differences, we also used the SF-36 health survey and the Knee Society Score as self-reported secondary outcomes (the latter includes a physical examination subscale).

ELIGIBILITY:
Inclusion Criteria:

* radiographically assessed osteoarthritis of the knee graded 1 to 4 according to the Kellgren and Lawrence scale
* self reported moderate to severe level pain

Exclusion Criteria:

* acute septic arthritis
* predisposition to a tendency to fall
* lack of physical or mental ability to perform or comply with the treatment procedure
* diabetes mellitus
* history of pathological osteoporotic fracture

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index (WOMAC)
Aggregated Locomotor Function (ALF)

SECONDARY OUTCOMES:
SF-36 health survey
Knee Society Score

CONTACTS AND LOCATIONS:
Overall Officials: Nahum Halperin, MD, Principal Investigator — Asaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Bar-Ziv Y, Beer Y, Ran Y, Benedict S, Halperin N. A treatment applying a biomechanical device to the feet of patients with knee osteoarthritis results in reduced pain and improved function: a prospective controlled study. BMC Musculoskelet Disord. 2010 Aug 10;11:179. doi: 10.1186/1471-2474-11-179. PMID 20698991